CLINICAL TRIAL: NCT00472537
Title: Prospective Randomized Evaluation of Open vs. Laparoscopic Operation of Ventral Incisional Eventrations. A Swedish Multicenter Study
Brief Title: ProLOVE - Prospective Randomized Study of Midline Incisional Hernia Treatment
Acronym: ProLOVE
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Region Skåne FoUU (Unknown); Lund University (Other); Ethicon, Inc. (Industry); The Einar & Inga Nilsson Foundation (Other); The Anna-Lisa & Sven-Eric Lundgren Foundation, Malmö Sweden (Other); Crafoord Foundation (Other)
Responsible Party: Principal Investigator, Peder Rogmark, M.D.,, Skane University Hospital
Other Study IDs: LU030123PR; 200-06-005
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: HERNIA, VENTRAL
Keywords: Ventral hernia; Incisional hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Retromuscular Mesh repair of midline incisional hernia
Procedure: Laparoscopic repair of midline incisional hernia

SUMMARY:
This purpose of this study is to compare the recovery after an operation of an incisional hernia within the limits of the rectus muscles of the abdominal wall. The use of a mesh in the repair of a postoperative hernia is considered obligatory. Placement of a retromuscular mesh is done by open or laparoscopic surgery. Focus is on the recovery phase assuming a less painful recovery after a laparoscopic procedure.

DETAILED DESCRIPTION:
Incisional ventral hernia after abdominal surgery is a fairly common condition. In recent years the use of a prosthesis in the repair procedure has proved very effective in preventing a new hernia. A retromuscular mesh placement seems to have superior results. The mesh may be placed retromuscular through an open surgical procedure or through a laparoscopic procedure in an intra-abdominal position. Both procedures are highly standardized. A heavy weight mesh is used in the open procedure, fixed in the midline only, and a composite mesh is used intraabdominally and fixed only with titanium tackers.

SF-36 is used to assess the quality of life, and its subscale BP (bodily pain) is used as primary outcome 3 weeks postoperatively. Secondary endpoints are return to daily life, pain, complications, recurrence, patient satisfaction and cosmetic outcome.

Subjects are assessed at 1,3,8 weeks post operation and after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Postoperative hernias in the region of the recti abdomini muscles with a defect of less than 10 cm transversal width
* No contraindications to laparoscopic procedure
* The patient should be able to adequate ventilation/respiration after reduction of hernia contents
* Indications for elective surgery

Exclusion Criteria:

* Pregnant women
* Prior operation of abdominal hernia with mesh placement in the compartment of the rectus abdominus muscle (i.e. prior onlay mesh is acceptable)
* Need of an interpreter
* Current drug abuse, mental disorder or other condition which makes the patient incapable of postoperative follow up
* Body Mass index (BMI) >40
* Other planned concurrent operation
* Current oral steroid treatment, or other immune system modulating treatment
* Incarcerated incisional hernias
* Parastomal hernias
* Prior history of open abdomen
* Enterocutaneous fistula or cutaneous infection
* Hepatic cirrhosis or ascites
* Generalized malignancy
* History of radiation treatment in the abdomen.
* ASA >III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to specialist centers for treatment of midline incisional hernias.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2005-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pain recorded in SF-36 | 3 weeks after surgery
  Pain measured 3 weeks after surgery in SF36 subscale Bodily Pain

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Montgomery, MD, PhD, Principal Investigator — Malmo University Hospital, Lund University
Locations (7):
- Sweden (7):
  - Malmö University Hospital, Department of Surgery, Malmo, Malmö
  - Arvika Hospital, Department of Surgery, Arvika
  - Helsingborg Hospital, Department of Surgery, Helsingborg
  - Lund University Hospital, Department of Surgery, Lund
  - Mora Hospital, Department of Surgery, Mora
  - Södertälje Hospital, Department of Surgery, Södertälje
  - Västerås Central Hospital, Department of Surgery, Västerås

REFERENCES:
- [Derived] Rogmark P, Ekberg O, Montgomery A. Long-term retromuscular and intraperitoneal mesh size changes within a randomized controlled trial on incisional hernia repair, including a review of the literature. Hernia. 2017 Oct;21(5):687-696. doi: 10.1007/s10029-017-1624-9. Epub 2017 Jun 20. PMID 28634690
- [Derived] Rogmark P, Petersson U, Bringman S, Eklund A, Ezra E, Sevonius D, Smedberg S, Osterberg J, Montgomery A. Short-term outcomes for open and laparoscopic midline incisional hernia repair: a randomized multicenter controlled trial: the ProLOVE (prospective randomized trial on open versus laparoscopic operation of ventral eventrations) trial. Ann Surg. 2013 Jul;258(1):37-45. doi: 10.1097/SLA.0b013e31828fe1b2. PMID 23629524